CLINICAL TRIAL: NCT04308369
Title: Follow-up of Osteo-articular Biomarkers After Spa Therapy at Dax in a Population With Knee Osteoarthritis and Their Correlation With the Clinical Evolution
Brief Title: Follow-up of Osteo-articular Biomarkers After Spa Therapy in a Population With Knee Osteoarthritis and Their Correlation With the Clinical Evolution
Acronym: BIOMARTHROSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ch Mont de Marsan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A02801-56
Record Dates: First submitted 2020-03-05; First posted 2020-03-16 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; spa therapy; osteo-articular markers
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: interventional study with minimal risk. Ony blood collection done during study to determinate biological marker level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood collection arm (Other): Blood collection will be performed before the spa therapy (Day 0), at the end of the spa therapy (Week 3) and 6 months later (M6).
  Interventions: Biological: Blood collection arm

INTERVENTIONS:
Biological: Blood collection arm — Blood collection will be performed before the spa therapy (Day 0), at the end of the spa therapy (Week 3) and 6 months later (M6). In this study, blood samples will be collected by a nurse of the service and centralized by the laboratory of Medical Biology of the General hospital of Dax.

SUMMARY:
Spa therapy is used in the treatment of various diseases and mainly osteoarthritis. Knee osteoarthritis is a very common rheumatic disease whose prevalence increases with longer life span and is a public health problem.

The Forestier and al. study highlighted the actual benefit and confirmed the improvement of the quality of life and pain of the knee osteoarthritis patients from 6 months of spa treatment.[1] A significant decrease of 30% in the rate of Serum Hyaluronic Acid at 6 months after the end of the spa therapy was also highlighted in the Canteloup et al study.[6] This study aims to measure different osteoarticular biomarkers (hyaluronic acid, coll2-1 and CTX1) before, at the end of the spa therapy and 6 months after the spa therapy and correlate with the clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with knee osteoarthritis defined according to the recommendations of the American College of Rheumatology (ACR):

  * painful articulation and at least one of the following three criteria: age > 50 years and/or articular crepitation and/or morning stiffness less than 30min
  * and radiographic sign of gonarthrosis with osteophyte (on X-rays of less than 3 years).
* Patient can come to the final visit at 6 months and living within a perimeter of 30km around Dax.
* Patient affiliated to a social security scheme.

Exclusion Criteria:

* Osteoarthritis limited to patellofemoral joint.
* A previous spa therapy of less than 6 months.
* Spa therapies with double indication rheumatology and phlebology.
* Patient with osteoporosis.
* A known hepatocellular failure or known acute or end-stage renal failure.
* Severe depressive syndrome, psychotic syndrome, immune deficiency, cardiopathy, evolutive neoplasia or infection.
* Infiltration and/or viscosupplementation < 6 months.
* Change in anti-osteoarthritis treatment of less than 3 months.
* Patient under tutorship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Describe the change of serum level of Hyaluronic acid (a marker of synovial inflammation) | 6 months (timepoint: at Day 0, Week 3 and month 6)
  Measure of serum level of Hyaluronic acid before the spa therapy (Day 0), at the end of the spa therapy (Week 3) and 6 months later (M6).

SECONDARY OUTCOMES:
Marker of cartilage degradation: Coll2-1 | 6 months (timepoint: at Day 0, Week 3 and month 6)
  Measure of biological marker of cartilage degradation (Coll2-1) before the spa therapy (Day 0), at the end of the spa therapy (Week 3) and 6 months later (M6).
Marker of bone resorption: CTX1 | 6 months (timepoint: at Day 0, Week 3 and month 6)
  Measure of biological marker of bone resorption (CTX1) before the spa therapy (Day 0), at the end of the spa therapy (Week 3) and 6 months later (M6).
Index of symptomatic severity of knee osteoarthritis or WOMAC | 6 months (timepoint: at Day 0, Week 3 and month 6)
  Patients will have been asked to answer symptom questionnaire (WOMAC) before the spa therapy (Day 0), at the end of the spa therapy (Week 3) and 6 months later (M6). It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items), Stiffness (2 items) and Physical Function (17 items). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.
Pain evaluation Visual Analogue Scale | 6 months (timepoint: at Day 0, Week 3 and month 6)
  Patients will have been asked to answer pain questionnaire (EVA) before the spa therapy (Day 0), at the end of the spa therapy (Week 3) and 6 months later (M6). The EVA is in the form of a 10 cm plastic strip graduated in mm. On the face presented to the patient, there is a cursor which he mobilizes along a straight line, one end of which corresponds to "No pain", and the other to "Maximum pain imaginable". The patient must, along this line, position the cursor at the place that best locates his pain. On the other side, there are millimeter graduations seen only by the caregiver. The position of the cursor mobilized by the patient makes it possible to read the intensity of the pain, which is measured in mm.
SF 36 Quality of Life Questionnaire | 6 months (timepoint: at Day 0, Week 3 and month 6)
  Patients will have been asked to answer and quality of life questionnaire (SF-36) before the spa therapy (Day 0), at the end of the spa therapy (Week 3) and 6 months later (M6). There are 11 questions in SF-36, with 36 items in total.
  The SF-36 items are divided into 8 different areas: Physical component (4 areas: Physical activity, Limitations due to physical condition, Physical pain, Perceived health) and Mental component (4 areas: Life and relationships with others , Psychic health, Limitations due to mental state, Vitality).
  It is requested to respond according to the last 4 weeks. The rating system recommended for the SF-36 is a weighted Likert system for each item. The items in the subscales are totaled in order to obtain a summary score for each subscale or dimension. Each of the 8 summary scores is linearly transformed on a scale of 0 (negative for health) to 100 (favorable for health) to obtain a score for each subscale.
Global clinical evaluation with kne flexion and joint swelling | 6 months (timepoint: at Day 0, Week 3 and month 6)
  A global clinical evaluation done with evaluation of different exams: Knee flexion (in degrees), joint swelling (measuring the perimeter of the joint (in cm)) before the spa therapy (Day 0), at the end of the spa therapy (Week 3) and 6 months later (M6).

CONTACTS AND LOCATIONS:
Overall Officials: Charles COWAN, MD, Principal Investigator — CH de Dax
Locations (1):
- centre hospitalier Dax, Dax, France

REFERENCES:
- [Result] Forestier R, Desfour H, Tessier JM, Francon A, Foote AM, Genty C, Rolland C, Roques CF, Bosson JL. Spa therapy in the treatment of knee osteoarthritis: a large randomised multicentre trial. Ann Rheum Dis. 2010 Apr;69(4):660-5. doi: 10.1136/ard.2009.113209. Epub 2009 Sep 3. PMID 19734131